CLINICAL TRIAL: NCT00673946
Title: Impact of Oximetry on Hospitalization
Brief Title: Impact of Oximetry on Hospitalization in Acute Bronchiolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Suzanne Schuh, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1000011675
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; hospitalization; oximetry; pediatrics
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): In this arm, patients are monitored with oximeters displaying true saturation values
  Interventions: Other: True saturation values displayed
- 2 (Experimental): In this arm, patients are monitored with oximeters with displayed saturations 3 percentage points above true values
  Interventions: Other: Altered saturation values displayed.

INTERVENTIONS:
Other: True saturation values displayed — Physicians will be presented with real saturations.
  Arms: 1
Other: Altered saturation values displayed. — Physicians will be presented with saturation measurements three percentage points above the true values.
  Arms: 2

SUMMARY:
To determine, in previously healthy infants 6 weeks to 12 months of age, diagnosed with acute bronchiolitis and monitored by hourly oximetry, if the probability of hospitalization within 72 hours of arrival in those whose oxygen saturation display is manipulated 3 percentage points above the true measurements is significantly lower in comparison to those whose monitors display true saturations.

DETAILED DESCRIPTION:
This is the first bronchiolitis study to examine the clinical and economic impact of making disposition decision on primarily clinical grounds, while blinding the physicians to oxygen saturations by providing them with either true saturation measurements or those which are 3 percentage points above the true values. Although physiologically insignificant and within the measurement error of the instrument, this difference has been shown to be perceived as clinically relevant and to have a major hypothetical impact on disposition, without any evidence to support this belief.

We hope to find out if children with oxygen saturations above or in the vicinity of the threshold recommended for initiation of oxygen therapy by the AAP can be safely discharged based on their clinical appearance rather than to have their hospitalization dictated by a locally defined number. This study will hopefully provide much needed evidence necessary to help us interpret the oximetry results more meaningful which may in turn lead to fewer hospitalizations, shorter length of hospital stay and lower health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Acute bronchiolitis
* Age 4 weeks to 12 months
* Baseline Respiratory Disease Assessment Instrument (RDAI) ≥ 3 points
* Informed consent
* Availability of a telephone

Exclusion Criteria:

* Pre-existing pulmonary or cardiac distress, neuromuscular disease, congenital or acquired airway anomalies, hemoglobinopathies, or chronic hypoxia
* Severe respiratory distress, defined as the retraction component on the RDAI as 8 out of possible 9 points
* True baseline oxygen saturation less than 88% in room air
* Transfers from other institutions

Ages: 6 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2008-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hospitalization for bronchiolitis | 72 hours from start of study

SECONDARY OUTCOMES:
The proportions of infants receiving supplemental oxygen in the ED | 72 hours from start the study
Length of stay in the ED (from the time of arrival to the disposition decision) | Determined by outcome measure
Proportions of infants with unscheduled medical visits for bronchiolitis symptoms to any medical facility | 72 hours from start of study.
Proportion of the ED staff/fellows in "strong agreement" or "agreement" with discharge | 0, 60, 120, 180, 240, 300, and 360 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Schuh, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Schuh S, Freedman S, Coates A, Allen U, Parkin PC, Stephens D, Ungar W, DaSilva Z, Willan AR. Effect of oximetry on hospitalization in bronchiolitis: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):712-8. doi: 10.1001/jama.2014.8637. PMID 25138332